CLINICAL TRIAL: NCT06309030
Title: Clinical Study on the Deep Remission of Rheumatoid Arthritis With Kidney Deficiency and Excessive Cold Syndrome by Bushen Quhan Zhiwang Decoction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Longxiao (Other)
Responsible Party: Sponsor-Investigator, Liu Longxiao, Doctor, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZRJY2023-QM21
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Drug: Bushen quhan zhiwang decoction
- Control group (Placebo Comparator)
  Interventions: Drug: Bushen quhan zhiwang decoction placebo

INTERVENTIONS:
Drug: Bushen quhan zhiwang decoction — Treatment with 100ml of Bushen quhan zhiwang decoction twice a day for 3 months.
  Arms: Intervention group
Drug: Bushen quhan zhiwang decoction placebo — Treatment with 100ml of Bushen quhan zhiwang decoction placebo twice a day for 3 months.
  Arms: Control group

SUMMARY:
The investigators conduct this randomized controlled clinical trial to evaluate the efficacy and safety of the Bushen Quhan Zhiwang decoction in patients with RA with kidney deficiency and excessive cold syndrome who have not achieved deep remission and remained at a low level of disease activity despite the use of conventional synthetic disease-modifying antirheumatic drugs.

DETAILED DESCRIPTION:
In this study, a randomized, double-blind, placebo-controlled clinical research methodology was proposed using computerized SPSS software to randomize the group to include 72 cases of RA patients who had been treated regularly with traditional RA disease-improving antirheumatic drugs for more than 3 months and whose disease was still at a low level of disease activity. On the basis of RA traditional condition-improving antirheumatic drug treatment, the treatment group was given Inib soup to tonify the kidney, dispel cold and cure the inibs, and the control group was given an analog of Inib soup to tonify the kidney, dispel cold and cure the inibs, with a 12-week treatment period and a 4-week follow-up period, in order to observe the efficacy and safety of the inibs based on the tonifying the kidney, dispel cold and cure the inibs on the clinical depth of relief of RA pain, and to assess the DAS-28, the VAS score of pain, the mechanical pain threshold, and laboratory laboratory laboratory tests (blood and urine routine, liver and renal function, ESR, CRP, RF, ACPA), electrocardiogram, compare the differences between the two groups in each of the above indexes and conduct correlation analysis, so as to provide evidence-based medical evidence for clinical practice. Based on clinical practice, explore the effect of tonifying the kidney, dispelling cold and curing Inibs to improve the clinical remission of RA, and provide a new strategy for the standardized treatment and clinical remission of RA. Using a combination of pain VAS scores and objective mechanical pain threshold measurements, we evaluated the effect of tonifying the kidneys, dispelling cold, and curing inibs on the pain relief of RA patients with kidney deficiency and cold-sheng syndrome, and provided references for the relief of RA pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting the ACR/European League against Rheumatism (EULAR) 2010 classification criteria；
2. Patients meeting the diagnostic crite ria (2018 edition) for "kidney deficiency and excessive cold syndrome" in Chinese medicine；
3. The disease activity score derivative for 28 joints (DAS28) score should be 2.6 to 3.2；
4. Use of traditional disease-modifying antirheumatic drugs (DMARDs), tretinoin preparations, etc., limited to 1 type and have been treated at a stable dose for at least 4 weeks prior to enrollment, and the dose of the medication remains unchanged after enrollment；
5. For those taking oral glucocorticosteroids prior to enrollment, the dose must be stabilized to a dose equivalent to ≤10 mg/day of prednisone for at least 4 weeks prior to enrollment and remain unchanged after enrollment；
6. Those using non-steroidal anti-inflammatory drugs (NSAIDs) or other analgesics for RA must have been on a stable dose for at least 1 week prior to enrollment and the dose of medication must remain unchanged after enrollment；
7. Voluntary participation and written informed consent.

Exclusion Criteria:

1. Previously treated with small molecule targeted drugs or biologics and discontinued for <4 weeks；
2. Those who have been treated with intra-articular, intramuscular or intravenous corticosteroids, including pro-adrenal hormones, within 4 weeks prior to enrollment；
3. Those with a combination of clearly diagnosed autoimmune diseases such as systemic lupus erythematosus, scleroderma, Sjogrensyndrome, etc.；
4. Organ transplant recipients, patients with malignant tumors, patients with heart, brain, liver (ALT/AST>3 times the upper limit of normal), kidney (Ccr<60ml/min) and other important organ function damage or blood system diseases；
5. With psychosomatic disorders such as cognitive impairment, depression, anxiety, and somatic dysfunction, central nervous disorders such as cerebral infarction, cerebral hemorrhage, epilepsy, TIA, myelitis, demyelinating lesions, or peripheral neurological disorders such as restless leg syndrome；
6. Women and men who are pregnant or breastfeeding or who plan to become pregnant in the next 6 months; women of childbearing age who are unable or unwilling to use adequate contraception or whose partners are unwilling to use contraception, either during the trial period or within 1 month after the last dose of medication；
7. BMI greater than 35 (kg/m2), allergic to the test drug, or participating in other clinical trials；
8. Other conditions deemed by the investigator to make participation in the trial unsuitable (out-of-town patients unable to follow up, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
disease activity score derivative for 28 joints (DAS28) | Enrolment, 4 weeks, 8 weeks,12 weeks and 16 weeks after intervention.
  DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96; DAS28 (ESR) = 0.56*√(TJC28)+0.28*√(SJC28)+0.014*GH+0.70*ln(ESR), where TJC = tender joint count and SJC = swollen joint count.

SECONDARY OUTCOMES:
patient reported outcomes（PRO） | Enrolment, 4 weeks, 8 weeks,12 weeks and 16 weeks after intervention.
  assessed by a dedicated rheumatologist (associate senior physician or better)
visual analogue scale for pain | Enrolment, 4 weeks, 8 weeks,12 weeks and 16 weeks after intervention.
  assessed by a dedicated rheumatologist (associate senior physician or better)
withdrawl mechanical threshold | Enrolment, 4 weeks, 8 weeks,12 weeks and 16 weeks after intervention.
  Von Frey test：The value of the minimum force that causes the patient to feel "pain" is the patient's mechanical pain threshold.
erythrocyte sedimentation Rate（ESR） | Enrolment, 4 weeks,12 weeks after intervention.
  Measured by the Laboratory of China-Japan Friendship Hospital
C-reactive protein（CRP） | Enrolment, 4 weeks,12 weeks after intervention.
  Measured by the Laboratory of China-Japan Friendship Hospital
TCM symptom score | Enrolment, 4 weeks, 8 weeks,12 weeks and 16 weeks after intervention.
  assessed by a dedicated rheumatologist (associate senior physician or better)